CLINICAL TRIAL: NCT03545425
Title: FoxBioNet: LRRK2-002: Detection of LRRK2 Activity in Human Biospecimens
Brief Title: Fox BioNet Project: LRRK2-002
Status: Completed | Type: Observational
Sponsor: Michael J. Fox Foundation for Parkinson's Research (Other)
Collaborators: University Health Network, Toronto (Other); Indiana University (Other); University of Rochester (Other)
Responsible Party: Principal Investigator, Connie Marras, Neurologist at Toronto Western Hospital Movement Disorders Centre, University Health Network, Toronto
Other Study IDs: LRRK2002
Record Dates: First submitted 2018-05-22; First posted 2018-06-04 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Biomarker; LRRK2
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Idiopathic Parkinson's Disease patients: Up to 30 Parkinson's Disease patients will be enrolled.
  Interventions: Procedure: Biofluid samplings
- Healthy Controls: Up to 30 Healthy Controls will be enrolled.
  Interventions: Procedure: Biofluid samplings
- LRRK2 G2019S - Manifesting: Up to 30 LRRK2 G2019S Manifesting carriers will be enrolled.
  Interventions: Procedure: Biofluid samplings
- LRRK2 G2019S - Non-Manifesting: Up to 30 LRRK2 G2019s Non-Manifesting carriers will be enrolled.
  Interventions: Procedure: Biofluid samplings

INTERVENTIONS:
Procedure: Biofluid samplings — Blood and Urine

SUMMARY:
The overall objective of this study is to determine whether LRRK2 kinase activity and/or mitochondrial DNA (mtDNA) damage could serve as potential biomarkers in PD.

DETAILED DESCRIPTION:
Primary Objectives:

* Assess the levels of phosphorylated LRRK2 and LRRK2-phosphorylated Rabs, as measures of LRRK2 kinase activity, in PBMCs and neutrophils from LRRK2 PD, idiopathic PD, non-manifesting LRRK2 mutation carriers and healthy controls.
* Assess the levels of mtDNA damage in buffy coat from LRRK2 PD, idiopathic PD, non-manifesting LRRK2 mutation carriers and healthy controls.
* Correlate LRRK2 kinase activity to mtDNA damage in blood from LRRK2 PD, idiopathic-PD, non-manifesting LRRK2 mutation carriers and healthy controls.

Secondary Objectives:

* To assess the ability of the network to efficiently conduct a study involving biosample collection for PD research. Efficiency will be assessed using measures of the time taken to meet specific milestones within the study.
* To assess the ability of the network to collect high quality biospecimens adhering to agreed-upon, standardized protocols
* To gauge the willingness of participants to participate in subsequent Fox BioNet studies

ELIGIBILITY:
Inclusion Criteria:

LRRK2 Parkinson Disease (PD) Subjects:

* Patients must have confirmed LRRK2 mutation
* Patients must meet the MDS criteria for Parkinson's disease
* Disease duration: any
* Male or female age 30 years or older at time of PD diagnosis.

Idiopathic PD Subjects:

* Patients must meet the MDS criteria for Parkinson's disease.
* Disease duration: any
* Male or female age 30 years or older at time of PD diagnosis.

Non-manifesting LRRK2 mutation carriers:

* Patients must have confirmed LRRK2 mutation
* Male or female age 30 years or older at Screening.

Control (C) Subjects:

* Male or female age 30 years or older at Screening.

Exclusion Criteria:

LRRK2 Parkinson Disease (PD) Subjects:

* Inability to provide informed consent
* Participation in a blinded clinical trial of any kind or an unblinded trial of an investigational product that is not currently approved for use in humans.
* Treatment for cancer in the last 5 years.

Idiopathic PD Subjects:

* Inability to provide informed consent
* Participation in a blinded clinical trial of any kind or an unblinded trial of an investigational product that is not currently approved for use in humans.
* Treatment for cancer in the last 5 years.

Non-manifesting LRRK2 mutation carriers:

* Inability to provide informed consent
* Participation in a blinded clinical trial of any kind or an unblinded trial of an investigational product that is not currently approved for use in humans.
* Treatment for cancer in the last 5 years.

Control Subjects:

* Inability to provide informed consent
* Participation in a blinded clinical trial of any kind or an unblinded trial of an investigational product that is not currently approved for use in humans.
* Treatment for cancer in the last 5 years

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 LRRK2 G2019S Manifesting carriers, 30 Idiopathic PD subjects, 30 LRRK2 G2019S Non-Manifesting Carriers, 30 Healthy Controls
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Phosphorylated LRRK2 and LRRK2-phosphorylated Rabs | 7 months
  Assess the levels of phosphorylated LRRK2 and LRRK2-phosphorylated Rabs, as measures of LRRK2 kinase activity, in PBMCs and neutrophils from LRRK2 PD, idiopathic PD, non-manifesting LRRK2 mutation carriers and healthy controls.
mtDNA damage in buffy coat | 7 months
  Assess the levels of mtDNA damage in buffy coat from LRRK2 PD, idiopathic PD, non-manifesting LRRK2 mutation carriers and healthy controls.
Correlate LRRK2 kinase activity to mtDNA damage | 7 months
  Correlate LRRK2 kinase activity to mtDNA damage in blood from LRRK2 PD, idiopathic-PD, non-manifesting LRRK2 mutation carriers and healthy controls.

SECONDARY OUTCOMES:
Assess the ability of the network to efficiently conduct a study | 7 months
  To assess the ability of the network to efficiently conduct a study involving biosample collection for PD research. Efficiency will be assessed using measures of the time taken to meet specific milestones within the study.
Assess the ability of the network to collect high quality biospecimens | 7 months
  To assess the ability of the network to collect high quality biospecimens adhering to agreed-upon, standardized protocols
To gauge the willingness of participants to participate in subsequent Fox BioNet studies | 7 Months
  To gauge the willingness of participants to participate in subsequent Fox BioNet studies

CONTACTS AND LOCATIONS:
Overall Officials: Connie Marras, MD, Principal Investigator — University Health Network, Toronto
Locations (5):
- United States (5):
  - Charles E. Schmidt College of Medicine, Florida Atlantic University, Boca Raton, Florida
  - Northwestern University, Chicago, Illinois
  - Columbia University Medical Center, New York, New York
  - Oregon Health and Sciences University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No